CLINICAL TRIAL: NCT06070467
Title: Holistic Mixed Approaches to Capture the Real Life of Children With Rare Eye Diseases
Acronym: SeeMyLife
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8826
Record Dates: First submitted 2023-09-26; First posted 2023-10-06 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Eye Diseases; Severe Loss of Vision; Blindness; Quality of Life
MeSH Terms: conditions — Eye Diseases; Vision Disorders; Blindness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children and teenagers affected by Rare Eye Diseases: A Mixed Methods Research (MMR) using quantitative (QUAN) Vision Related-QoL (VR-QoL = FVQ-CYP and VQoL-CYP) tools and psychosocial PEM-CY, and qualitative (QUAL) socio-anthropologic investigations can capture reliably children's and teenagers' Patient-Reported Outcome (PRO).
  Interventions: Other: Mixed Methods Research (MMR) using quantitative (QUAN) and qualitative (QUAL) tools

INTERVENTIONS:
Other: Mixed Methods Research (MMR) using quantitative (QUAN) and qualitative (QUAL) tools — A Mixed Methods Research (MMR) using quantitative (QUAN) Vision Related-QoL (VR-QoL = FVQ-CYP and VQoL-CYP) tools and psychosocial PEM-CY, and qualitative (QUAL) socio-anthropologic investigations can capture reliably children's and teenagers' Patient-Reported Outcome (PRO).
  The QUAN study is a cross-sectional study including short-term re-test repetition (children/teenagers only) using the following PROMs for children/teenagers:
  1. Self-reported questionnaires for patients (FVQ-CYP and VQoL-CYP)
  2. For caregivers: PEM-CY questionnaires
  The QUAL study will rely on the following instruments:
  1. Semi-directive interviews,
  2. Focus groups,
  3. Field observation.

SUMMARY:
Rare Eye Diseases (RED) are the leading cause of severe visual impairment/ blindness (SVI/B) in children in Europe. This sensory disability with its accompanying psychological distress hugely impacts their lives and their families. Understanding this impact, at a patient centred level, is key in care, in shared decision making, in developing therapies, and in improving social integration and participation about the standard rules of the United Nations (UN) and the European Union (EU) (prevention, non-discrimination, equal opportunities, accessibility, etc.). However, current tools to evaluate vision related (VR) quality of life (QoL) VR-QoL disregard age and cultural differences. There is a lack knowledge on how the disease matters at child's level. Instruments capable of yielding high-quality data, psychometrically robust and comply with regulatory requirements remain to be developed.

To fill this gap, SeeMyLife will use multilevel concurrent mixed method research combining quantitative studies and qualitative studies. The quantitative approach is based on (i) cross culturally translated validated VR-QoL questionnaires for children and teenagers (Functional Vision Questionnaire for Children and Young People - FVQ-CYP and Vision-related Quality of Life Questionnaire for Children and Young People - VQoL-CYP) and (ii) on caregiver's questionnaires addressing participation and environment (Participation and Environment Measure - Children and Youth - PEM-CY). To fully capture the picture of the child/teenager personal life the investigators will reinforce their investigations by in depth qualitative socio-anthropologic study with semi directive field interviews and fieldwork (to observe closely the living conditions of the children) to address how their impairment affects their wellbeing, social integration, and how they feel about medical and social interventions. Data analysis will use an integrated mixed method strategy to validate the quantitative tools and deliver a holistic QoL transnational tool.

The SeeMyLife project will provide (i) robust patient self-reported tools that will be then used in care and research (especially with the rise in novel therapies) as a standard as well as (ii) highly awaited knowledge about the SVI/B patient's position within his own life course, within his family and in relation to health and social care actors.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 8-12) and teenagers (age 13-18) with various levels of visual impairment defined according to World Health Organization (WHO) International Classification of Diseases (ICD) 10 - WHO ICD 10 [best-corrected visual acuity ≤ 0.3 decimal or ≤ 6/18], and their parents/caregivers.

Exclusion Criteria:

* Children, teenagers, and caregivers:

  1. who lack the ability to respond in a reliable way to the questions on how they feel about their visual impairment (patients with mild intellectual or cognitive deficiency may be able to reply accurately as opposed to cases with severe intellectual disability)
  2. with functional or non-ophthalmic reasons of visual impairment
  3. unable to provide consent/assent;
  4. who do not speak/read the language

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children (age 8-12) and teenagers (age 13-18) with various levels of visual impairment defined according to World Health Organization (WHO) International Classification of Diseases (ICD) 10 - WHO ICD 10 [best-corrected visual acuity ≤ 0.3 decimal or ≤ 6/18], and their parents/caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
real-life impact of SVI/B in children and teenagers affected by Rare Eye Diseases | 12 months
  To elucidate whether Patient-Reported Outcome Measures (PROMs) reflect how children/teenagers perceive their lives to be impacted by Rara Eye Diseases using Vision-related Quality of Life Questionnaire for Children and Young People - VQoL-CYP

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence pour les Affections Rares en Génétique Ophtalmologique (CARGO), Hôpitaux Universitaires, Strasbourg, France